CLINICAL TRIAL: NCT00491816
Title: Phase II Trial of Neoadjuvant Erlotinib Plus Chemotherapy for Treatment of ER Negative, PgR Negative and HER-2 Negative Primary Breast Cancer
Brief Title: Erlotinib Plus Chemotherapy for Treatment of Triple Negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10864
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: breast; cancer; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Erlotinib Hydrochloride; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- erlotinib with neoadjuvant chemotherapy (Experimental): Study drug, erlotinib, is administered along with neoadjuvant chemotherapy. Adjuvant therapy given at discretion of treating physician. Once adjuvant therapy is completed, all patients will receive erlotinib 150 mg daily for 1 year.
  Interventions: Drug: Erlotinib with neoadjuvant chemotherapy

INTERVENTIONS:
Drug: Erlotinib with neoadjuvant chemotherapy — 150 mg orally (PO) once daily on days 3 to 14, given with cycle 1 to 6 or 3 to 6 of neoadjuvant chemotherapy
  Other Names: Tarceva

SUMMARY:
Primary Study Objective:

To assess the pathological complete response rate (pCR) with 4-6 cycles of neoadjuvant chemotherapy plus erlotinib in patients with triple negative breast cancer.

DETAILED DESCRIPTION:
Twenty percent of women with breast cancer have triple negative breast cancer. The standard treatment for triple negative breast cancer is typically a combination of chemotherapy, surgery, +/- radiation therapy. When treated with standard therapy women with triple negative breast cancer have a worse long term outcomes as compared to women who do not have triple negative breast cancer. Triple negative breast cancer cells usually have a surface marker called EGFR (epidermal growth factor receptor). Women whose breast cancer cells have the EGFR surface marker have worse long term outcomes as compared to women whose tumors do not have the EGFR marker. Erlotinib (Tarceva) targets EGFR and is currently used for treatment of other cancers like lung and pancreas. This study will assess a combination of chemotherapy with erlotinib in women with triple negative breast cancer.

For breast cancer patients who receive chemotherapy first and then get surgery, long-term survival is longer for women who do not have any microscopic cancer at the time of surgery. The primary objective of this study is to assess whether a combination of chemotherapy and erlotinib will result in no evidence of microscopic disease (pCR) at the time of surgery in greater than 20% of enrolled subjects. After completing all chemotherapy, patients will also receive maintenance erlotinib for 12 months. This is given to study the tolerability of maintenance Erlotinib and also to evaluate if maintenance erlotinib will decrease the rate of tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Female patient ≥ 18 years of age
* Histologically proven stage II or III adenocarcinoma of the breast
* Patients must be candidates for neoadjuvant treatment (tumor size > 2 cm, T2, T3, T4 and/or clinical N1 or N2)
* Estrogen Receptor negative, Progesterone Receptor negative and HER-2 negative disease (IHC 0 or 1+ and/or FISH negative)
* Performance status of 2 or better
* No prior chemotherapy or endocrine therapy
* If female of childbearing potential, pregnancy test is negative and willing to use effective contraception while on treatment and for at least 3 months after the last dose of study drug
* Adequate bone marrow function: neutrophils ≥ 1500/mm3, platelet count ≥ 100,000/mm3, and hemoglobin ≥ 11 g/dL
* Adequate kidney function: serum creatinine ≤ 1.5 mg/dl and/or creatinine clearance of ≥ 60 mL/min
* Adequate hepatic function: transaminases < 2 x upper limit of normal and total bilirubin ≤ 1.5 mg/dL
* Patients must have a serum albumin ≥ 3.0 g/dL
* Patients must have a Prothrombin Time, Partial Thromboplastin Time within normal limits
* Patients must be informed of the investigational nature of the study, and must sign an informed consent in accordance with the institutional rules
* Pretreatment lab values must be performed within 14 days of patient registration, and other baseline studies within 30 days
* Patients will have a baseline mammogram, bone scan, CT chest and abdomen

Exclusion Criteria:

* Patients with metastatic disease are excluded from study
* The presence of any other medical or psychiatric disorder that, in the opinion of the treating physician, would contraindicate the use of drugs in this protocol or place the subject at undue risk for treatment complications
* Pregnancy or lactation
* Prior use of an Epidermal growth factor receptor inhibitor
* Patients with a history of chronic pulmonary disease are excluded from study
* Patients with inadequate laboratory values (as defined above) are excluded from study
* Patients with NCI common toxicity criteria (CTC) grade 2 or greater peripheral neuropathy are excluded from study
* Patients with active infection are excluded from study
* Patients with concomitant or previous malignancies within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, are excluded from study
* Patients with emotional limitations are excluded from study
* Patients with inflammatory breast cancer will be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-07; Primary Completion 2014-12 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | After 18 weeks of neoadjuvant therapy

SECONDARY OUTCOMES:
Estimation of change in ki-67 (proliferation) after 2 cycles of neoadjuvant carboplatin/docetaxel based chemotherapy | After 2 cycles (6 weeks) of therapy
Estimation of change in ki-67 after 2 cycles of carboplatin/docetaxel based neoadjuvant chemotherapy plus erlotinib | After 2 cycles (6 weeks) of therapy
Assessment of toxicity of the combination of carboplatin/docetaxel chemotherapy plus erlotinib | During neoadjuvant chemotherapy
Assessment of tolerability of 12 months of maintenance erlotinib treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka Sharma, M.D., Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States